CLINICAL TRIAL: NCT03312322
Title: Effects of Lumbar Transcutaneous Electrical Nerve Stimulation on Exercise Performance in Patients With Chronic Obstructive Pulmonary Disease : A Pilot Study
Brief Title: Effects of Lumbar Transcutaneous Electrical Nerve Stimulation on Exercise Performance in Patients With Chronic Obstructive Pulmonary Disease
Acronym: LENS-REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LENS-REHAB
Record Dates: First submitted 2017-09-27; First posted 2017-10-17 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Three constant workload testing will be performed on three different days.
  Every test will be carried out with a different condition :
  * Sham transcutaneous electrical nerve stimulation;
  * High-frequency transcutaneous electrical nerve stimulation;
  * Low-frequency transcutaneous electrical nerve stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham placebo will be used to blind patient. The outcome assessor will be invited to join the room after the experimental condition is installed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CWT with high-frequency electrical nerve stimulation (Experimental): This study has a cross-over design. Patients will achieve CWT with either sham, high-frequency or low-frequency lumbar transcutaneous electrical nerve stimulation in a randomised order.
  Interventions: Other: High-frequency transcutaneous electrical nerve stimulation
- CWT with low-frequency electrical nerve stimulation (Experimental): This study has a cross-over design. Patients will achieve CWT with either sham, high-frequency or low-frequency lumbar transcutaneous electrical nerve stimulation in a randomised order.
  Interventions: Other: Low-frequency transcutaneous electrical nerve stimulation
- CWT with sham electrical nerve stimulation (Experimental): This study has a cross-over design. Patients will achieve CWT with either sham, high-frequency or low-frequency lumbar transcutaneous electrical nerve stimulation in a randomised order.
  Interventions: Other: Sham transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: High-frequency transcutaneous electrical nerve stimulation — 4 self adhesive surface electrodes are positioned by pair at the L3-L4 level, laterally.
  Stimulation is setted at rest, 10min before constant workload testing. During this period, intensity is increased every 3minutes to the maximum tolerated by the patient (pain threshold). Thereafter, intensity is not increased anymore during the test.
  It is explained to the patient that he might or no experience the electrical stimulation sensation.
  Current characteristics : 100Hertz, 100ms, bidirectional. Constant workload testing : 60-70rpm ; 75% Wpic ; up to exhaustion or rpm < 60 during more than 10s.
  Arms: CWT with high-frequency electrical nerve stimulation
Other: Low-frequency transcutaneous electrical nerve stimulation — 4 self adhesive surface electrodes are positioned by pair at the L3-L4 level, laterally.
  Stimulation is setted at rest, 10min before constant workload testing. During this period, intensity is increased every 3minutes to the maximum tolerated by the patient (pain threshold). Thereafter, intensity is not increased anymore during the test.
  It is explained to the patient that he might or no experience the electrical stimulation sensation.
  Current characteristics : 4Hertz, 100ms, bidirectional. Constant workload testing : 60-70rpm ; 75% Wpic ; up to exhaustion or rpm < 60 during more than 10s.
  Arms: CWT with low-frequency electrical nerve stimulation
Other: Sham transcutaneous electrical nerve stimulation — The procedure is the same as high-frequency transcutaneous electrical stimulation but intensity is progressively setted back to 1mA (over a 45sec period) after every increment so that constant workload testing is performed with 1mA.
  Arms: CWT with sham electrical nerve stimulation

SUMMARY:
Chronic obstructive pulmonary disease is a leading cause of morbidity and mortality worldwide.

Pulmonary rehabilitation effectively improves outcomes in patients with chronic respiratory disease. There is a link between training intensity and physiological improvements following pulmonary rehabilitation. However, high intensity training is not sustainable for every patients.

Therefore, actual strategies for pulmonary rehabilitation aimed at decreasing dyspnea to improve muscle work.

Electrical muscle stimulation is widely used during rehabilitation to promote muscle function recovery. Transcutaneous electrical nerve stimulation was recently used to relief dyspnea and improve pulmonary function in patients with chronic respiratory disease. Moreover, spinal anesthesia with fentanyl has been shown to be effective in improving exercise tolerance in patients with chronic obstructive pulmonary disease (inhibiting group III and IV muscle afferents). As transcutaneous electrical muscle stimulation stimulates the same receptors in the spinal cord dorsal horn as fentanyl, it is hypothesized that it could also improve exercise capacity.

Therefore, the aim of this study is to assess wether transcutaneous electrical stimulation (high or low frequency) is effective in improving exercise capacity in patients with severe to very severe chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Design : cross-over.

Patients will perform three constant workload testing (CWT) on different days under three different conditions. The intervention during the tests will be randomly assigned (concealed allocation) :

* Sham transcutaneous electrical nerve stimulation ;
* High-frequency transcutaneous electrical nerve stimulation ;
* Low-frequency transcutaneous electrical nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Chronic obstructive pulmonary disease Gold III-IV;
* Eligible for pulmonary rehabilitation;
* Never used electrical stimulation.

Non-inclusion Criteria:

* Pregnant woman or likely to be;
* Patient under guardianship;
* History of epilepsy, heart pace-maker or defibrillator, inguinal or abdominal hernia;
* Recent lumbar surgery or skin lesion;
* Allergy to surface electrodes;
* Lumbar sensitivity impairment;
* Opiate treatment during the last 3 months.

Exclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Comparison of endurance time (Tlim, in second) during constant workload testing (CWT) under 3 conditions. | The outcome will be measured after every CWT. Data will be continuously collected during the tests. The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
  Patients will achieve 3 constant workload testing under 3 different conditions (sham lumbar transcutaneous electrical nerve stimulation, high-frequency lumbar electrical nerve stimulation and low-frequency lumbar transcutaneous electrical nerve stimulation). Endurance time (sec) will be recorded at the end of every test. Endurance time will be compared to assess how the condition will influence exercice performance.

SECONDARY OUTCOMES:
Dyspnea during CWT using modified Borg Scale (0-10). | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be collected every 30s during tests
  The dyspnea will be assessed every 30sec during CWT. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Exhaustion during CWT using modified Borg Scale (0-10). | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be collected every 30s during tests.]
  The exhaustion will be assessed every 30sec during CWT. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Heart rate (rpm) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Blood pressure (mmHg) before and after every CWT. | The outcome will be assessed before and after every CWT. The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum.
Oxygen saturation (SpO2, %) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
O2 consumption (VO2, mL/kg/min) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Exercise ventilation (VE, L/min) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Tidal Volume (Vt, L) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Respiratory Rate (RR, rpm) during CWT. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Variation of total hemoglobin (THb) using near infra red spectroscopy. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Variation of total desoxy-hemoglobin (HHb) using near infra red spectroscopy. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Variation of total oxy-hemoglobin (HbO2) using near infra red spectroscopy. | The outcome will be measured during every CWT.The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected
  Outcome will be continuously recorded. Results will be shown at Tlim (Tlim for the 3 tests) and iso time (defined as the Tlim or the shortest test).
Intensity of electrical stimulation (mA) reached during every CWT. | The outcome will be measured after every CWT. The 3 CWT will be carried out in different days, separate from 1 day minimum for a total time frame of 2 weeks maximum. Data will be continuously collected

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuvelier, Prof, PhD, Principal Investigator — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Catherine Tardif, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Catherine Viacroze, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; David Debeaumont, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Maxime Patout, MD, MsC, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Lamia Bouchra, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, PT, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Tristan Bonnevie, PT, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, France

IPD SHARING:
Plan to Share IPD: Undecided